CLINICAL TRIAL: NCT05891977
Title: Development of Sustainable Tomato Products to Improve the Microbiota-gut-brain Axis: From Farm to Fork to Health (MITOS)
Brief Title: Effect of Tomato Paste Consumption on the Microbiota-gut-brain Axis in Healthy Adults
Acronym: MITOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Rosa M Lamuela-Raventós, Professor, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PID2020-114022RB-I00
Record Dates: First submitted 2023-05-17; First posted 2023-06-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-02

CONDITIONS: Microbiota; Cognitive Function; Healthy Lifestyle
Keywords: Carotenoid; Inflammation Mediators; Preventive Medicine; Polyphenols; Tomato; Clinical trial

STUDY DESIGN:
Intervention Model Description: Intervention A: Habitual diet + consumption of low to moderate tomato or tomato products and other food sources of lycopene + 0.5 g of tomato paste / kg of body weight (experimental intervention) for 3 months.
  Intervention B: Habitual diet + consumption of low to moderate tomato or tomato products and other food sources of lycopene (control) for 3 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group AB (intervention / control) (Experimental): After a 1-week washout period avoiding consumption of tomato, tomato-based products and other food sources of lycopene (watermelon, papaya, grapefruit and lycopene supplements), participants will consume a daily amount of 0.5 g of tomato paste / kg of body weight following the regular diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods during 3 months (intervention). Then they will return to their regular dietary pattern during 3 weeks. At the beginning of the first 4 month, participants will be encouraged to move into the second phase (control), before a 1-week washout period. The second phase or control consists in following their regular diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods during the next 3 months.
  Interventions: Other: Intervention A - Tomato paste; Other: Intervention B - Control
- Group BA (control / intervention) (Experimental): After a 1-week washout period avoiding consumption of tomato, tomato-based products and other food sources of lycopene (watermelon, papaya, grapefruit, and lycopene supplements), participants will start the control intervention which consists of following their regular diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods during 3 months (control). Then they will return to their regular diet during 3 weeks. At the beginning of the first 4 month, participants will be encouraged to move into the second phase (intervention), before a 1-week washout period. The intervention consist in consuming a daily amount of 0.5 g of tomato paste / kg of body weight diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods during the next 3 months.
  Interventions: Other: Intervention A - Tomato paste; Other: Intervention B - Control

INTERVENTIONS:
Other: Intervention A - Tomato paste — Participants will consume a daily amount of 0.5 g of tomato paste / kg of body weight following the regular diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods
Other: Intervention B - Control — Participants will consume the regular diet plus consumption of low to moderate tomato or tomato-based products and lycopene containing foods

SUMMARY:
Tomatoes and tomato-based products could play an important role in modulating microbiota-gut-brain axis (MGBA) interactions due to their high content of fiber and phytochemicals. Phytochemical metabolites derived from the consumption of tomato-based products can act directly as neurotransmitters in the central nervous system, crossing the blood-brain barrier, or indirectly by modulating the MGBA. These metabolites can thus alter gut bacterial composition and brain biochemistry. Therefore, researchers propose a new interventional study to assess the impact of daily tomato consumption in the organism, and to evaluate the effect on the MGBA. The final aim of this study is to spread a message of the health benefits of tomato consumption for the general population.

DETAILED DESCRIPTION:
To evaluate the possible changes in microbiota and cognitive skills after consumption of tomato paste in a crossover randomized controlled study. Fifty healthy adults subjects (aged 40-55 years and consisting of 50% males and 50% females to assess possible sex-based responses) will be included. Participants will sign the informed consent and carry out a washout period without consuming any tomatoes or tomato-based products during 1 week. Participants will consume a daily amount of 0.5 g of tomato paste / kg of body weight following the regular diet plus consumption of low to moderate tomato or tomato-based products and other sources of lycopene (experimental intervention), and the normal diet plus consumption of low to moderate tomato or tomato-based products and other sources of lycopene (control intervention) during 3 months. Biological samples (plasma, peripheral blood mononuclear cells, serum, 24-hours urine, feces, and saliva) will be obtained at baseline and the end of each arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects with BMI < 30 kg/m2
* Signed informed consent

Exclusion Criteria:

* Participants with tomato allergy or intolerance
* Cardiovascular disease (cancer or diabetes)
* Mental disorders (e.g. depression, dementia, autism, etc.)
* Cardiovascular alterations in triglycerides or glucose
* Participants with body mass index (BMI) > 30 kg/m2
* Current smokers
* Frequent use of corticoids, nonsteroidal anti-inflammatory drugs
* Volunteers with extreme eating habits (i.e. Atkins diet, very high protein diets, etc.)
* Excessive alcohol consumption (>30 g/d for males and >20 g/d for females),
* Pregnant or lactating women

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Changes in brain-derived neurotrophic factor (BDNF) after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Serum samples will be analysed for mature BDNF using a Mature BDNF Rapid ELISA kit.
Changes in cognitive function (executive) after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  The Wisconsin Sorting Cards Test (WSCT) will assess strategic planning, organized searching, utilizing environmental feedback to shift cognitive sets, directing behaviour towards achieving a goal and modulating impulsive responding.
Changes in cognitive function (attention) after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  The d2 Test will meausure selective and sustained attention and visual scanning speed. Processing speed, rule compliance, and quality of performance will be assess in participants.
Changes in cognitive function (memory) after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  The face-name associative memory exam (FNAME) will assess associative memory function.Participants will be asked to remember a set of faces and the names they are paired with. After a 5-25 minute delay, participants will recall which of the faces and names they saw earlier.
Changes in cerebrovascular function after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Cerebrovascular function will be measured using functional magnetic resonance imaging (FMRI), a non-invasive method for assessing brain activity. FMRI maps blood oxygenation levels in the brain and estimates changes in the blood flow that depends on metabolic function and is correlated with specific brain region activities
Changes in the gut microbiota after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Fecal samples will be collected by the volunteers using a system for easy self-collection and stabilization of microbial DNA for gut microbiome profiling (OMNIgene - GUT). The genomic DNA will be extracted from fecal samples using the DNeasy PowerSoil Kit. Then, microbial profiling using 16S ribosomal RNA (rRNA) sequencing will be used to study microbial communities, specially bacterial phylogeny and taxonomy.
Changes in the polyphenols and carotenoids and their metabolites after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Carotenoids and polyphenols, and their metabolites derived from intestinal gut microbiota will be identified and quantified in human plasma, urine, feces, and saliva samples using High Performance Liquid Chromatography HPLC-LTQ-Orbitrap-MS/MS and HPLC-MS/MS techniques.
Changes in the short-chain fatty acids in plasma and feces samples after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  After acidifying the fecal samples with formic acid, a quantification of short-chain fatty acids will be performed using gas chromatography by direct injection according to previously described methodology (Zhao et al., 2006).
Changes in bile acids in plasma and feces samples after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Bile acids will be assayed using a validated liquid chromatography-mass spectrometry (LC-MS) method

SECONDARY OUTCOMES:
Changes in Body mass index after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Body mass index (kg/m^2) will be calculated after measuring weight (kg) and height (meters).
Changes in waist-to-hip ratio with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Waist and hip circumferences (cm) will be measured in triplicate and then combined to report waist-to-hip ratio.
Changes in anthropometric measurements after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Body mass index (kg/m^2) will be calculated after measure weight (kg) and height (meters). To evaluate waist-to-hip ratio, waist and hip circumferences (cm) will be measured in triplicate.
Changes in body composition after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Body fat percentage will be measured using a bioelectrical impedance analysis monitor.
Changes in blood pressure after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Diastolic and systolic blood pressure will be measured by a blood pressure monitor in triplicate.
Changes in heart rate after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Heart rate (bpm) will be measured with an automatic monitor in triplicate.
Changes in lipidic profile after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (mg/dL) will be measured by molecular absorption spectrometry.
Changes in liver function after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP) and albumin will be assayed by immunoenzymatic methods.
Changes in glucose after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Glucose (mg/dL) will be measured by molecular absorption spectrometry.
Changes in pro- and anti-inflammatory biomarkers after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Cytokines (pg/mL), tumor necrosis factor α (TNF-α) (pg/mL) and C-reactive protein (CRP) (mg/dL) will be assayed by immunoenzymatic methods.
Changes in nutrients and energy intake after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  A 7-day food recall will be used. The data will be analyzed using a software called Programa de Càlcul Nutricional Professional (PCN Pro).
Changes in quality of the diet after each intervention with tomato paste and the control intervention. | Baseline
  Participants will fill the validated questionnaire measuring adherence to the Mediterranean diet.
Changes in physical activity after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Physical activity will be assessed with the ActiGraph® wGT3X-BT accelerometer.
Changes in sleep quality after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Sleep quality will be assessed with the ActiGraph® wGT3X-BT accelerometer.
Changes in quality of life after each intervention with tomato paste and the control intervention. | Baseline and after completed each intervention (3 months)
  Quality of life will be assessed with the WHOQOL-BREF.
Sensory threshold and organoleptic analysis | Baseline
  The recognition threshold of the five basic tastes will be determined through a classical sensory analysis test, employing a battery of solutions containing the molecules of interest. This test will include an organoleptic analysis of tomato paste to evaluate its aroma, taste (including acidity, sweetness, saltiness, umami), and hedonic sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa M Lamuela Raventós, PhD, Principal Investigator — University of Barcelona
Locations (1):
- Department of Nutrition, Food Sciences and Gastronomy. School of Farmacy and Food Sciences. University of Barcelona., Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No